CLINICAL TRIAL: NCT07160309
Title: Effect of Densah Bur Versus Magnetic Mallet Device on Osseodensification of Narrow Alveolar Ridge for Implant Placement
Brief Title: Osseodensification and Ridge Expansion for Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Reham Abdelrahman, assistant lecturer at OMFs Department - Deraya University, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-SU-22-02
Record Dates: First submitted 2025-08-15; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Alveolar Bone Loss
Keywords: Osseodensification Dental Implants
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Densah Bur (Experimental): Participants in this arm will undergo implant site preparation using the Densah bur system for osseo
  Interventions: Device: Densah Bur
- Magnetic Mallet (Experimental): Participants in this arm will undergo implant site preparation using the Magnetic Mallet device for
  Interventions: Device: Magnetic Mallet

INTERVENTIONS:
Device: Densah Bur — Implant site preparation will be performed using the Densah bur system to achieve osseodensification in narrow alveolar ridges prior to implant placement.
  Arms: Densah Bur
Device: Magnetic Mallet — Implant site preparation will be performed using the Magnetic Mallet device to achieve osseodensification in narrow alveolar ridges prior to implant placement.
  Arms: Magnetic Mallet

SUMMARY:
Ridge expansion techniques allow implant placement in narrow alveolar ridges by increasing bone volume using the native bone. This technique has shown to be a safe and effective procedure.

DETAILED DESCRIPTION:
This clinical study aims to evaluate the effectiveness of ridge expansion techniques in patients with narrow alveolar ridges characterized by low bone density. The procedure relies on using the patient's native bone to increase ridge volume, allowing for successful placement of dental implants without the need for extensive grafting. The study will compare different expansion methods in terms of bone gain, implant stability, and complication rates. By assessing clinical and radiographic outcomes, the trial seeks to determine the predictability and safety of ridge expansion as a minimally invasive alternative for implant site development.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with partial edentulous alveolar ridges with adequate alveolar bone height and deficient width and density.
2. Patients with good state of health and free from systemic or local pathosis that may influence the outcome of the therapy.
3. Good oral hygiene.
4. Age above 18 years.
5. Agreement to participate in the study and also have to be able to attend postoperative clinical and radiological follow-up schedule.

Exclusion Criteria:

1. Patients with para-functional habits such as bruxism and clenching or abnormal occlusal relationship that may complicate the future restoration.
2. Patients with bad oral hygiene or smokers.
3. Patients with uncontrolled systemic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Title: Primary Implant Stability (ISQ Values) | Time Frame: At the time of implant placement (Day 0).
  Description: Measurement of implant stability quotient (ISQ) using resonance frequency analysis immediately after implant placement.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Mohamed, Phd, Principal Investigator — Al-Azhar University
Locations (1):
- Faculty of Dentistry, Department of Oral and Maxillofacial Surgery, Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT07160309/Prot_000.pdf